CLINICAL TRIAL: NCT01364974
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential Group, Multiple-Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ASP015K in Healthy, Non-Elderly Male and Female Adult Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 015K-CL-HV02
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP015K; Pharmacodynamics
Keywords: ASP015K; Healthy subjects
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Experimental): low dose, all male
  Interventions: Drug: ASP015K; Drug: Placebo
- Group B (Experimental): medium dose, all male
  Interventions: Drug: ASP015K; Drug: Placebo
- Group C (Experimental): high dose, all male
  Interventions: Drug: ASP015K; Drug: Placebo
- Group D (Experimental): medium dose, all female
  Interventions: Drug: ASP015K; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP015K — oral
  Arms: Group A; Group B; Group C; Group D
Drug: Placebo — oral

SUMMARY:
The objective of this study is to explore safety and tolerability of multiple oral doses of ASP015K in healthy volunteers.

DETAILED DESCRIPTION:
Subjects will be confined to the clinical research unit for 19 days. Subjects will receive a follow-up phone call to asses safety 1 to 5 days after being discharged from the study.

Subjects will receive study drug twice per day (BID) on days 1 to 13 of the 14 day treatment period, and will receive a single dose of study drug on the morning of day 14 of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* If female, the subject is at least 2 years post menopausal or is surgically sterile per documentation provided by a third party medical professional and the subject is not pregnant as documented by a negative serum pregnancy test
* If male, the subject agrees to sexual abstinence and/or to use a highly effective method of birth control during the study period
* Subject is medically healthy, with no clinically significant abnormalities on medical history or abnormalities observed upon physical examination or 12 lead electrocardiogram (ECG)
* Subject's fasting clinical laboratory values are within normal limits
* Subject is a non-smoker or a light smoker (< 10 cigarettes/day)
* Subjects must weigh at least 45 kg and have a Body Mass Index (BMI) of 18-32 kg/m2

Exclusion Criteria:

* Subject has a positive test for hepatitis C antibody, or positive for hepatitis B surface antigen (HBsAg)
* Subject is known positive for human immunodeficiency virus (HIV) antibody
* Subject has a history of severe allergic or anaphylactic reactions
* Subject has a history of chronic diarrhea
* Subject has been vaccinated within the last 60 days prior to study drug administration
* Subject has a previous history of any clinically significant neurological, gastrointestinal, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the Investigator's opinion, would preclude participation in the study
* Subject has had clinically significant illness within 1 month prior to study drug administration
* Subject has a history of hemorrhoids
* Subject has a positive guaiac test
* Subject has a history of drug or alcohol abuse, a positive urine or serum screen for drugs of abuse/illegal drugs, or positive blood or breathalyzer for alcohol
* Subject has had treatment with prescription medication (except hormone replacement therapy and acetaminophen), complementary and alternative medicines (CAM) within 14 days, over-the-counter products within 1 week, or alcohol, caffeine or grapefruit juice within 24 hours prior to study drug administration
* Subject has had treatment with another investigational drug or approved therapy for investigational use within 30 days or 10 half-lives, whichever is longer, prior to study drug administration or has participated in a prior group in the current study
* Subject has a history of blood donation within 30 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed through vital signs, electrocardiograms (ECGs), physical exams, reports of adverse events, and analysis of blood and urine samples | 25 days
Pharmacokinetic assessment through the analysis of blood and urine samples | 17 days
Pharmacodynamic assessment through the analysis of blood samples | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States